CLINICAL TRIAL: NCT06207656
Title: Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of Cetuximab in Combination with Encorafenib Plus Binimetinib As Induction Treatment in BRAF V600E Mutated MSS Initially Resectable or Potentially Resectable Advanced Colorectal Cancer
Brief Title: Study to Evaluate the Efficacy and Safety of Cetuximab in Combination with Encorafenib Plus Binimetinib As Induction Treatment in BRAF V600E Mutated MSS Initially Resectable or Potentially Resectable Advanced Colorectal Cancer
Acronym: CEBBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Merck, S.L., Spain (Industry); Pierre Fabre Ibérica, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-21-02
Record Dates: First submitted 2023-12-27; First posted 2024-01-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer
Keywords: BRAF V600E mutated; MSS; advanced colorectal cancer; Cetuximab; Encorafenib; Binimetinib
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cetuximab in combination with encorafenib plus binimetinib (EBC) (Experimental): Patients will receive the following per 28-day cycle:
  * Encorafenib: 300 mg (4 × 75 mg oral capsule) daily (QD)
  * Binimetinib: 45 mg (3 × 15 mg oral tablet) twice daily (BID)
  * Cetuximab: 500 mg/m2 every 2 weeks as per standard institutional practice.
  Interventions: Drug: EBC

INTERVENTIONS:
Drug: EBC — Patients will receive the following per 28-day cycle:
  * Encorafenib: 300 mg (4 × 75 mg oral capsule) daily (QD)
  * Binimetinib: 45 mg (3 × 15 mg oral tablet) twice daily (BID)
  * Cetuximab: 500 mg/m2 every 2 weeks as per standard institutional practice.

SUMMARY:
As a result of the little benefit obtained from standard treatments and the poor prognosis of these patients, the BRAF-V600E mutant MSS aCRC represents an unmet medical need requiring clinical research.

The combination of encorafenib, cetuximab and binimetinib as second- or third-line treatment for mCRC resulted in significantly better outcomes than standard therapy in a phase 3 clinical trial, which also revealed treatment safety and tolerability to be acceptable. Compared to the control group (cetuximab and irinotecan or cetuximab and FOLFIRI), the triplet therapy cohort showed higher median overall survival (9.3 vs. 5.9 months) and response rates (26.8% vs. 1.8%). Grade 3 adverse events occurred in 65.8% and 64.2% of patients for triple-therapy and control groups, respectively.

Based on these results, the investigators speculated that the combination of encorafenib, cetuximab and binimetinib could be used as induction therapy to improve treatment outcomes in BRAF-V600E-mutated MSS aCRC locally advanced initially unresectable but potentially resectable; initially resectable or initially unresectable but potentially resectable oligometastatic disease; and in patients with stage II-IV who have relapsed after chemotherapy (neo and/or adjuvant) or surgery, if the shorter time after resection or from treatment end to relapse is longer than 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female participants age ≥18 years at the time of informed consent. 2. Capable of giving signed informed consent/assent. 3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

  4. Participants with histologically or cytologically confirmed colorectal adenocarcinoma.

  5. Presence of a BRAF V600E mutation confirmed as per standard of care according to international guidelines at any time prior to Screening.

  6. Microsatellite stable (MSS) or Mismatch-Repair proficient (pMMR) disease confirmation assessed by local PCR or immunohistochemistry (IHC).

  7. Participants with CRC who have one of these criteria:
  1. Locally advanced colorectal cancer with initially unresectable but potentially resectable disease according to the local Multidisciplinary Tumour Board (MTB).
  2. Oligometastatic colorectal cancer (possible metastasis sites: liver, lung, lymph nodes and peritoneum) with:

  i. Initially resectable disease according to the local MTB or ii. Initially unresectable but potentially resectable disease according to the local MTB c. Stage II-IV colorectal cancer treated with previous neoadjuvant and/or adjuvant chemotherapy, for R0, if the shorter time from the resection or from the end of the adjuvant treatment to the relapse of colorectal cancer (possible metastasis sites: liver, lung, lymph nodes and peritoneum) is longer than 6 months. This relapse (locoregional and/or systemic) should be initially resectable or initially unresectable but potentially resectable disease according to the local MTB 8. ECOG performance status of 0 or 1. 9. Measurable or evaluable disease as assessed by investigator, according to RECIST v1.1.

  10. Adequate bone marrow function characterized by the following at screening:
  1. ANC ≥1.5 × 109/L
  2. Platelets ≥100 × 109/L
  3. Hemoglobin ≥9.0 g/dL (with or without blood transfusions). 11. Adequate hepatic and renal function characterized by the following at screening:

  <!-- -->

  1. Serum total bilirubin ≤1.5 x ULN. Note 1: Total bilirubin >1.5 x ULN is allowed if direct (conjugated) ≤1.5 x ULN and indirect (unconjugated) bilirubin is ≤4.25 x ULN.

     Note 2: Participants with hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the medical monitor.
  2. ALT and AST ≤2.5 × ULN, or ≤5 × ULN in the presence of liver metastases.
  3. Adequate renal function defined by an estimated creatinine clearance ≥50 mL/min according to the Cockcroft Gault formula or by 24-hour urine collection for creatinine clearance, or according to local institutional standard method.

     12. Able to swallow, retain, and absorb oral medications.

     Exclusion Criteria:
* 1. Any medical or psychiatric condition including recent (within the past year) or current suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

  2. Leptomeningeal disease or brain metastases. 3. History of chronic inflammatory bowel disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to the start of study treatment.

  4. Known RAS-mutant colorectal adenocarcinoma. 5. Impaired gastrointestinal function (e.g., uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, small bowel resection) or disease which may significantly alter the absorption of oral study intervention or recent changes in bowel function suggesting current or impending bowel obstruction.

  6. Clinically significant cardiovascular diseases, including any of the following:
  1. History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) ≤6 months prior to the start of study treatment.
  2. Congestive heart failure requiring treatment (New York Heart Association Grade ≥2).
  3. History or presence of clinically significant cardiac arrhythmias (including uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia).
  4. History of thromboembolic or cerebrovascular events ≤12 weeks prior to the start of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e., massive or sub-massive) deep vein thrombosis or pulmonary emboli.

     Note 1: Participants with either deep vein thrombosis or pulmonary emboli that do not result in hemodynamic instability are allowed to enroll as long as they have been on a stable dose of anticoagulants for at least 4 weeks.

     Note 2: Participants with thromboembolic events related to indwelling catheters (including PICC lines) or other procedures may be enrolled.
  5. Triplicate average QTcF interval ≥480 ms or a history of prolonged QT syndrome.
  6. Congenital LQTS. 7. Evidence of active non-infectious pneumonitis. 8. Evidence of active and uncontrolled bacterial or viral infection, with certain exceptions, as noted below, for chronic infection with HIV, hepatitis B or hepatitis C (please see below), within 2 weeks prior to start of study treatment.

     9. Participants positive for HIV are ineligible unless they meet all of the following:

  <!-- -->

  1. A stable regimen of highly active anti-retroviral therapy that is not contraindicated.
  2. No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections.
  3. A CD4 count >250 cells/mcL, and an undetectable HIV viral load on standard PCR-based tests.

     10. Active hepatitis B or hepatitis C infection

  a. Active HBV is defined as any of the following:
  1. HBsAg (+), HBV DNA >200 IU/mL (105 copies/mL);
  2. HBsAg (+), HBV DNA ≤200 IU/mL and persistent or intermittent elevation of ALT/AST and/or liver biopsy showing chronic hepatitis with moderate or severe necroinflammation.

     Note: Participants who are HBsAg (-), HBcAb (+) are eligible and should be monitored/treated as per local standard of care.

  b. Active HCV is defined as:
  1. HCV antibody positive; AND
  2. Presence of HCV RNA. 11. Concurrent or previous other malignancy within 3 years of study entry, except curatively treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, Bowen's disease or prostate cancer with a Gleason score ≤6. Participants with other curatively treated malignancies with low risk of recurrence not listed may also be considered eligible after review and approval by the medical monitor.

     12. Residual CTCAE≥ Grade 2 toxicity from any prior anticancer therapy, with the exception of Grade 2 alopecia or Grade 2 neuropathy.

     13. Previous treatment with any selective BRAF inhibitor (e.g., encorafenib, dabrafenib, vemurafenib, XL281/BMS-908662) and/or any selective MEK inhibitor prior to screening.

     14. Use of any prohibited medication (including herbal medication), supplement or food that is a moderate or strong inhibitor or inducer of CYP3A4/5 ≤1 week prior to the start of study intervention.

     15. Major surgery (e.g., inpatient procedure with regional or general anesthesia) or completion of radiation therapy ≤4 weeks prior to the start of study treatment.

     16. Previous systemic anticancer therapy for CRC, with the following exceptions:

     • Patients with resected (R0 or R1 resections) metastasis of CRC treated with or without adjuvant or neoadjuvant chemotherapy (+/- antiEGFR or bevacizumab) would be includible if the time from the resection or from the end of the adjuvant treatment (the later) to the relapse of CRC were longer than 6 months

     • Patients with previous adjuvant or neoadjuvant chemotherapy for resected St II/III CRC would be eligible if the time from the resection or from the end of the adjuvant treatment (the later) to the relapse of CRC were longer than 6 months 17. Prior systemic regimen in first line treatment for metastatic CRC in patients with unresectable or non-potentially resectable metastatic (M1) disease.

     18. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

     19. Known contraindication to receiving cetuximab including hypersensitivity or toxicity that would suggest an inability to tolerate maximum cetuximab dose of 500 mg/m2.

     20. Known sensitivity or contraindication to any component of study intervention or their excipients at the planned doses.

     21. Pregnant, or is breastfeeding (lactating). 22. Male or female of childbearing age who do not agree with taking highly effective contraceptive precautions, (for definition, please refer to Appendix 15) or abstinence during the course of the study and for 6 months after the last administration of study drug for women and men.

     23. Full dose radiotherapy <28 days prior to the start of study treatment. Short course radiotherapy for local control of primary tumor or other palliative indication is allowed.

     24. Patients with ulcerative keratitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of cetuximab in combination with encorafenib plus binimetinib as induction therapy for the treatment of BRAF-V600E mutated MSS aCRC to perform radical treatment of the primary and/or metastases | From first dose to radical treatment (up 60 months)
  Radical treatment rate, defined as the number of patients radically treated for their primary tumor and/or distant metastases by surgery and/or by any other radical therapeutic procedure with curative intent (i.e. radiofrequency, cryotherapy, laserhyperthermia, stereotactic body radiotherapy or chemoembolization).

SECONDARY OUTCOMES:
Overall response rate (ORR) | From first dose to radiographic evidence of best response (up 60 months)
  Number of patients achieving complete response (CR) or partial response (PR) as best response according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, divided by the total number of patients.
Tumor regression grade (TRG), after any surgical treatment of the primary tumor and/or distant metastases | From surgery until 30 days post surgery (up 60 months)
  TRG1, no residual tumor; TRG2, microscopic residual tumor; TRG3, moderate response; TRG4, minor response; and TRG5, no response
Progression-free-survival (PFS) | From first dose to the earliest documented PD or death due to any cause (up 60 months)
  Time in months from first dose of study treatment to disease progression or death (due to any cause)
Overall survival (OS) | From first dose to death due to any cause (up 60 months)
  Time in months from first dose of study treatment to death due to any cause
Disease free survival (DFS) | From first dose to radiographic evidence of cancer recurrence, second cancer, or death (up 60 months)
  Time in months from first dose of study treatment to cancer recurrence, second cancer, or death from any cause in resected patients
Complications related to surgery and/or any other therapeutic procedure for radical treatment occurring within 60 days after surgery | From surgery until 30 days post surgery (up 60 months)
  Number of Participants with Perioperative mortality, transfusions, hemorrhage, infections, wound healing, general or local complications
Incidence and severity of AEs CTCAE v5 criteria | From first dose until 30 days post last dose of study treatment (up 60 months)
  Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and serious Adverse Events.

OTHER OUTCOMES:
To determine the presence/expression level/levels of serum and tumour tissue biomarkers associated with cell and tumour growth and/or involved in the mechanisms of action of EBC | Tumour tissue samples: at baseline and blood samples at baseline, at week12 post treatment and at progression
  To be confirmed

CONTACTS AND LOCATIONS:
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided